CLINICAL TRIAL: NCT00261118
Title: Phase 3: Randomised Controlled Trial of Rituximab in Active Ulcerative Colitis
Brief Title: Rituximab in Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal Liverpool University Hospital (Other Government)
Collaborators: Hoffmann-La Roche (Industry); University of Liverpool (Other)
Responsible Party: Principal Investigator, Jonathan Michael Rhodes, Invesitgator, Royal Liverpool University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLBUHT R&D 2709; DDX exemption from MRHA ref:-; MF 8000/12794
Record Dates: First submitted 2005-11-29; First posted 2005-12-02 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Ulcerative Colitis
Keywords: colitis; rituximab
MeSH Terms: conditions — Colitis, Ulcerative; Colitis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (i) (Active Comparator): Rituximab 1g in 500 mls of 0.9% normal saline infused into a peripheral vein
  Interventions: Drug: Rituximab
- 2 (ii) (Placebo Comparator): 500 mls of 0.9% NORMAL SALINE INFUSED INTO A PERIPHERAL VEIN
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 1g in 500 mls Normal Saline Placebo 500 mls Normal Saline
  Other Names: MabThera (Roche)

SUMMARY:
There is broad support for the hypothesis that Ulcerative colitis is an auto-immune disease. Rituximab is an antibody protein that removes a subgroup of white blood cells (B lymphocytes) from the circulation. These cells have the capacity to generate the auto-antibodies that typify auto-immune disease. Although Rituximab has been mainly used for treating B lymphocyte malignancies (lymphoma) it has also been used with promising results in Rheumatoid arthritis and has an excellent safety record. This is a small placebo-controlled trial to assess its efficacy and safety in patients with steroid-resistant active ulcerative colitis.

DETAILED DESCRIPTION:
WHAT IS THE PROBLEM TO BE ADDRESSED ?

Lack of effective cure for Ulcerative colitis.

WHAT IS THE HYPOTHESIS TO BE TESTED?

That rituximab may be effective in active ulcerative colitis.

WHY IS A TRIAL NEEDED NOW?

Rituximab has been used to treat more than 300,000 patients with B lymphocyte malignancies and has been shown to have an excellent safety record [6-8]. Published pilot studies have shown excellent results with rituximab in patients with autoimmune diseases such as immune-mediated thrombocytopaenia, Wegeners granulomatosis, cold agglutinin disease, myasthenia gravis, rheumatoid arthritis and SLE [11-17]. Together with increasing evidence to support a pathogenic role for the pANCA associated with ulcerative colitis, a study of rituximab in ulcerative colitis is timely. Moreover the only significant advance in the treatment of ulcerative colitis in recent years has been the introduction of cyclosporin which probably halves the colectomy rate [18,19] but at the risk of considerable side effects and with a drug-related mortality that has been estimated at 2%.

HAS A SYSTEMATIC REVIEW BEEN CARRIED OUT AND WHAT WERE THE FINDINGS?

A Medline search for " rituximab and ulcerative colitis" yielded no responses. There has been a recent report of its use in a single patient with ileocolonic Crohn's disease who also had immune-mediated thrombocytopaenia [20]. The thrombocytopaenia improved but the Crohn's disease did not. It can be argued though that there is little or no evidence for autoimmunity in Crohn's disease which seems in many cases to be due to a defect in phagocyte function, eg in association with the recently described NOD2/CARD15 genetic alteration.

2.5 HOW WILL THE RESULTS OF THIS TRIAL BE USED? This trial will establish whether rituximab is effective in achieving remission in patients with ulcerative colitis who are failing to respond to conventional therapy with corticosteroids. Because there is no background evidence of its efficacy the initial study will be a small two centre study with placebo blinding. If the result of this study is promising, these would be used as pilot data for power calculations for a larger multicentre study.

3.1 WHAT IS THE PROPOSED TRIAL DESIGN? A "placebo-blinded" study with 16 patients receiving rituximab and 6 patients receiving placebo (0.9% saline).

3.2 WHAT ARE THE PLANNED TRIAL INTERVENTIONS? Patients will receive either (i) rituximab 1g in 500 mls of 0.9% saline infused into a peripheral vein over four hours (see appended infusion chart), or (ii) 500 mls of 0.9% saline infused into a peripheral vein over two hours as placebo. This regimen will be repeated once at 2 weeks. This protocol is based on the dosing regimen that proved most efficacious for rheumatoid arthritis. All patients will also receive paracetamol 1g orally and chlorpheniramine (Piriton) 10mg intravenously immediately prior to each Rituximab/placebo infusion.

All patients will continue to receive oral prednisolone 40mg/day for 2 weeks then 30mg for two weeks, then 20mgs/day for two weeks, then reduce by 5mg/day every 7 days until off prednisolone.

3.3 WHAT IS THE PROPOSED DURATION OF THE TREATMENT PERIOD? Two treatments, two weeks apart.

3.4 WHAT ARE THE PROPOSED INCLUSION/EXCLUSION CRITERIA? see earlier

3.5 WHAT ARE THE PROPOSED OUTCOME MEASURES? see earlier 3.6 WILL HEALTH SERVICE RESEARCH ISSUES BE ADDRESSED? Not Applicable 3.7 WHAT IS THE PROPOSED FREQUENCY/DURATION OF FOLLOW UP? Patients will be reviewed after one, two and four, eight, twelve and twenty four weeks. Patients will be monitored thereafter in routine gastroenterology clinic follow up.

3.8 HOW WILL THE OUTCOME MEASURES BE MEASURED AT FOLLOW-UP? Patients will complete a daily diary with details of bowel frequency, presence of blood in the stool, any change in medical therapy and any new or worsening symptoms The IBD quality of life questionnaire will be completed at baseline and at weeks 4 and 12.

Patients will also have a diary card to record the details of any other symptoms noted during the trial to assess adverse effects of the trial treatment.

3.9 WHAT ARE THE PROPOSED PRACTICAL ARRANGEMENTS FOR ALLOCATING PATIENTS TO TRIAL GROUPS? Randomization will be allocated in blocks of five by the pharmacy department of the hospital.

3.10 WHAT ARE THE PROPOSED METHODS FOR PROTECTING AGAINST OTHER SOURCES OF BIAS? Controls (known only to the Pharmacy Department) will receive a placebo saline infusion.

3.11 WHAT IS THE PROPOSED SAMPLE SIZE? A "placebo-blinded" study with 16 patients receiving rituximab and 8 patients receiving placebo (0.9% saline). This will provide 80% power for excluding an 80% remission rate with active treatment compared with an assumed 25% placebo response.

3.12 WHAT IS THE PLANNED RECRUITMENT RATE? 1-2 patients per month 3.13 ARE THERE LIKELY TO BE ANY PROBLEMS WITH COMPLIANCE? No.

3.14 WHAT IS THE LIKELY RATE OF LOSS TO FOLLOW UP? 100% follow up should be achievable. 3.15 HOW MANY CENTRES WILL BE INVOLVED? Two 3.16 WHAT IS THE PROPOSED TYPE OF ANALYSIS? Formal hypothesis testing of the primary outcome will be compared by chi-square test.

Wilcoxon signed rank test will be used for comparisons against baseline for changes in secondary quantitative endpoints.

3.17 WHAT IS THE PROPOSED FREQUENCY OF ANALYSIS? Once only on completion. 3.18 ARE THERE ANY PLANNED SUBGROUP ANALYSES? Subgroup analysis may be performed according to pANCA status.

3.19 WHAT IS THE ESTIMATED RESEARCH COST OF THE TRIAL? Cost of therapy plus £800 pharmacy fee plus £2200 towards ethics submission/ research nurse time/ cost of pANCA assays to be provided as an unrestricted educational grant from Roche UK.

3.20 IS THERE AN NHS SERVICE SUPPORT COST OF THIS TRIAL, AND IF SO WHAT IS THE ESTIMATED COST? The only NHS cost would be modest, involving only the routine testing of full blood count and SMAC which is current practice in the monitoring of patients with relapses of inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over age of 18 years who are capable of providing written informed consent.
2. Confirmed diagnosis of ulcerative colitis by conventional clinical, endoscopic and histological criteria.
3. Failure of response to at least two weeks of oral prednisolone 40mg/day.
4. Active colitis as assessed by a Mayo score [21] of 6-12 inclusive (see Appendix 1)

Exclusion Criteria:

1. Patients under 18 or unable to give informed consent.
2. Patients in their first attack of ulcerative colitis.
3. Patients with severe ulcerative colitis as defined by presence of any of: temperature >37.5oC, pulse rate >100, focal severe or rebound abdominal tenderness, haemoglobin < 10.0g/dl, serum albumin <3.5 g/dl, transverse colon diameter greater than 5.0cms on plain abdominal X ray.
4. Patients who are pregnant, post partum (<3months) or breast feeding
5. Patients who are at risk of pregnancy and not using a reliable form of contraception (oral contraceptive and barrier or barrier plus spermicide).
6. Patients with a stoma
7. Positive stool culture for pathogens or test for C difficile at screening within 7 days prior to trial entry
8. Patients for whom a baseline Mayo score can not be reliably calculated: frequent use of laxatives (for proximal constipation) or antimotility agents (for control of diarrhoea)
9. Any change to maintenance medication for ulcerative colitis: azathioprine or 6-mercaptopurine within previous 3 months or 5-aminosalicylates within previous one month
10. Any change to rectal therapy for colitis within the previous two weeks.
11. Participation in other trials in the last 3 months.
12. Serious intercurrent infection or other clinically important active disease (including renal and hepatic disease)

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-04; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Remission defined as a decrease in Mayo score to ≤ 2 points at week 4 | week 4

SECONDARY OUTCOMES:
Clinical response defined as a decrease in Mayo score by ≥ 3 points at weeks 4, 8 (partial Mayo score) and 12. | Week 4, 8 & 12
Remission at weeks 8 and 12. | week 8 &12
Endoscopic mucosal healing at week 4 and 12 | Week 4 & 12
Improvement in Inflammatory Bowel Disease specific Quality of Life Index at weeks 4 and 12 | weeks 4 &12
Histological improvement of disease activity at 4 and 12 weeks compared with baseline. | week 4 & 12 weeks
Treatment tolerability as defined by adverse events. | all visits

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Rhodes, MD, Principal Investigator — University of Liverpool
Locations (1):
- Royal Liverpool University Hospital, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Background] Quinton JF, Sendid B, Reumaux D, Duthilleul P, Cortot A, Grandbastien B, Charrier G, Targan SR, Colombel JF, Poulain D. Anti-Saccharomyces cerevisiae mannan antibodies combined with antineutrophil cytoplasmic autoantibodies in inflammatory bowel disease: prevalence and diagnostic role. Gut. 1998 Jun;42(6):788-91. doi: 10.1136/gut.42.6.788. PMID 9691915
- [Background] Xiao H, Heeringa P, Hu P, Liu Z, Zhao M, Aratani Y, Maeda N, Falk RJ, Jennette JC. Antineutrophil cytoplasmic autoantibodies specific for myeloperoxidase cause glomerulonephritis and vasculitis in mice. J Clin Invest. 2002 Oct;110(7):955-63. doi: 10.1172/JCI15918. PMID 12370273
- [Background] Inoue N, Watanabe M, Sato T, Okazawa A, Yamazaki M, Kanai T, Ogata H, Iwao Y, Ishii H, Hibi T. Restricted V(H) gene usage in lamina propria B cells producing anticolon antibody from patients with ulcerative colitis. Gastroenterology. 2001 Jul;121(1):15-23. doi: 10.1053/gast.2001.25477. PMID 11438490
- [Background] Hibi T, Ohara M, Kobayashi K, Brown WR, Toda K, Takaishi H, Hosoda Y, Hayashi A, Iwao Y, Watanabe M, et al. Enzyme linked immunosorbent assay (ELISA) and immunoprecipitation studies on anti-goblet cell antibody using a mucin producing cell line in patients with inflammatory bowel disease. Gut. 1994 Feb;35(2):224-30. doi: 10.1136/gut.35.2.224. PMID 8307474
- [Background] Monteleone I, Vavassori P, Biancone L, Monteleone G, Pallone F. Immunoregulation in the gut: success and failures in human disease. Gut. 2002 May;50 Suppl 3(Suppl 3):III60-4. doi: 10.1136/gut.50.suppl_3.iii60. PMID 11953335
- [Background] Maloney DG, Liles TM, Czerwinski DK, Waldichuk C, Rosenberg J, Grillo-Lopez A, Levy R. Phase I clinical trial using escalating single-dose infusion of chimeric anti-CD20 monoclonal antibody (IDEC-C2B8) in patients with recurrent B-cell lymphoma. Blood. 1994 Oct 15;84(8):2457-66. PMID 7522629
- [Background] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Leandro MJ, Edwards JC, Cambridge G. Clinical outcome in 22 patients with rheumatoid arthritis treated with B lymphocyte depletion. Ann Rheum Dis. 2002 Oct;61(10):883-8. doi: 10.1136/ard.61.10.883. PMID 12228157
- [Background] De Vita S, Zaja F, Sacco S, De Candia A, Fanin R, Ferraccioli G. Efficacy of selective B cell blockade in the treatment of rheumatoid arthritis: evidence for a pathogenetic role of B cells. Arthritis Rheum. 2002 Aug;46(8):2029-33. doi: 10.1002/art.10467. PMID 12209504
- [Background] Arzoo K, Sadeghi S, Liebman HA. Treatment of refractory antibody mediated autoimmune disorders with an anti-CD20 monoclonal antibody (rituximab). Ann Rheum Dis. 2002 Oct;61(10):922-4. doi: 10.1136/ard.61.10.922. PMID 12228164
- [Background] Looney RJ. Treating human autoimmune disease by depleting B cells. Ann Rheum Dis. 2002 Oct;61(10):863-6. doi: 10.1136/ard.61.10.863. No abstract available. PMID 12228152
- [Background] Stasi R, Pagano A, Stipa E, Amadori S. Rituximab chimeric anti-CD20 monoclonal antibody treatment for adults with chronic idiopathic thrombocytopenic purpura. Blood. 2001 Aug 15;98(4):952-7. doi: 10.1182/blood.v98.4.952. PMID 11493438
- [Background] Specks U, Fervenza FC, McDonald TJ, Hogan MC. Response of Wegener's granulomatosis to anti-CD20 chimeric monoclonal antibody therapy. Arthritis Rheum. 2001 Dec;44(12):2836-40. doi: 10.1002/1529-0131(200112)44:123.0.co;2-w. PMID 11762944
- [Background] Patel DD. B cell-ablative therapy for the treatment of autoimmune diseases. Arthritis Rheum. 2002 Aug;46(8):1984-5. doi: 10.1002/art.10476. No abstract available. PMID 12209499
- [Background] Remuzzi G, Chiurchiu C, Abbate M, Brusegan V, Bontempelli M, Ruggenenti P. Rituximab for idiopathic membranous nephropathy. Lancet. 2002 Sep 21;360(9337):923-4. doi: 10.1016/S0140-6736(02)11042-7. PMID 12354476
- [Background] Leandro MJ, Edwards JC, Cambridge G, Ehrenstein MR, Isenberg DA. An open study of B lymphocyte depletion in systemic lupus erythematosus. Arthritis Rheum. 2002 Oct;46(10):2673-7. doi: 10.1002/art.10541. PMID 12384926
- [Background] Cohen RD, Stein R, Hanauer SB. Intravenous cyclosporin in ulcerative colitis: a five-year experience. Am J Gastroenterol. 1999 Jun;94(6):1587-92. doi: 10.1111/j.1572-0241.1999.01149.x. PMID 10364029
- [Background] Stack WA, Long RG, Hawkey CJ. Short- and long-term outcome of patients treated with cyclosporin for severe acute ulcerative colitis. Aliment Pharmacol Ther. 1998 Oct;12(10):973-8. doi: 10.1046/j.1365-2036.1998.00396.x. PMID 9798801
- [Background] Papadakis KA, Rosenbloom B, Targan SR. Anti-CD2O chimeric monoclonal antibody (rituximab) treatment of immune-mediated thrombocytopenia associated with Crohn's disease. Gastroenterology. 2003 Feb;124(2):583. doi: 10.1053/gast.2003.50081. No abstract available. PMID 12557172
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Guyatt G, Mitchell A, Irvine EJ, Singer J, Williams N, Goodacre R, Tompkins C. A new measure of health status for clinical trials in inflammatory bowel disease. Gastroenterology. 1989 Mar;96(3):804-10. PMID 2644154
- [Derived] Leiper K, Martin K, Ellis A, Subramanian S, Watson AJ, Christmas SE, Howarth D, Campbell F, Rhodes JM. Randomised placebo-controlled trial of rituximab (anti-CD20) in active ulcerative colitis. Gut. 2011 Nov;60(11):1520-6. doi: 10.1136/gut.2010.225482. Epub 2011 Apr 6. PMID 21471566